CLINICAL TRIAL: NCT02362009
Title: South Miami Hospital Fibroid Registry
Status: Terminated | Type: Observational
Why Stopped: Policy approved describing all procedures as standard of care
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Jaime Sepulveda, MD, Baptist Health South Florida
Other Study IDs: 13-099
Record Dates: First submitted 2015-01-20; First posted 2015-02-12 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Uterine Myomas, Leiomyomas, or Fibromas
Keywords: Myomas; Leiomyomas; Fibromas
MeSH Terms: conditions — Leiomyoma; Fibroma; Myoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the Fibroid Registry is to provide a comprehensive database that captures patient characteristics, clinical outcomes and pot-treatment quality of life measures for patients treated for uterine fibroids. This database will serve as a platform for future comparative effectiveness and other health services research studies.

DETAILED DESCRIPTION:
The proposed research will be a prospective registry study of patients treated for uterine fibroids at the Fibroid Center located at South Miami Hospitals Center for Women and Infants.

Our objective is to establish the Fibroid Registry:

* To collect and review short, middle and long term clinical outcomes data that will help inform and facilitate the decision making process of clinicians and patients on the safest and most effective treatment for symptomatic uterine myomas, leiomyomas, or fibromas.
* To be able to critically evaluate the quality of procedures being performed and to ultimately establish a gold standard of care based upon patient and clinical outcomes and characteristics.
* To ultimately establish a gold standard of care based upon clinical outcomes and patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seeking treatment for uterine myomas, leiomyomas, or fibromas.
2. Patients between the ages of 18-89.
3. Patients that agree to participate and sign consent.

Exclusion Criteria:

1)Patients that decline to participate and/or are younger than 18 or older than 89.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients seen for fibroid treatment services.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Short, middle and long term clinical outcomes data that will help inform and facilitate the decision making process of clinicians and patients on the safest and most effective treatment for symptomatic uterine myomas, leiomyomas, or fibromas. | Data elements will be collected at baseline prior procedure, at follow up for 30 days (± 5 days), 6 months (±5 days) and 12 months (± 5 days) post procedure.

SECONDARY OUTCOMES:
Critically evaluate quality of procedures being performed and ultimately establish a gold standard of care based upon patient, clinical outcomes and characteristics (Fibroid Questionnaire & Quality of Life Questionnaire) | Baseline prior procedure, at follow up for 30 days (± 5 days), 6 months (±5 days) and 12 months (± 5 days) post procedure.
  Such registry will enable us to address a number of research questions, for instance:
  * Is uterine artery embolization (UAE) a safe treatment for leiomyomata?
  * Is UAE an effective treatment for leiomyomata?
  * What is the likelihood of symptom relief?
  * How durable is the treatment?
  * What is the likelihood that a woman who undergoes UAE and plans subsequent pregnancy will be able to conceive and deliver a subsequent intrauterine pregnancy?
  * Are women choosing this procedure content with their selection?
  * Are there certain patient subgroups at higher risk or that have an increased likelihood of treatment benefits?

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Sepulveda, M.D, Principal Investigator — Principal Investigator
Locations (1):
- South Miami Hospital, Miami, Florida, United States